CLINICAL TRIAL: NCT01855620
Title: The Effect of Body Mass Index on Etonogestrel Levels in Women Using the Single-rod Contraceptive Implant
Brief Title: The Effect of Body Mass Index on Etonogestrel Hormone Levels in Women Using the Single-rod Contraceptive Implant
Acronym: Eto BMI
Status: Completed | Type: Observational
Sponsor: Columbia University (Other)
Responsible Party: Principal Investigator, Kathleen M. Morrell, Assistant Professor of Clinical Obgyn, Columbia University
Other Study IDs: AAAK6606
Record Dates: First submitted 2013-05-14; First posted 2013-05-16 (Estimated); Last update posted 2014-04-14 (Estimated); Status verified 2014-04

CONDITIONS: Contraception; Obesity
Keywords: Contraception; Implant; Obesity
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole blood
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Normal weight women: Women with implant for more than twelve months who have BMI <25.
- Overweight women: Women with implant for more than twelve months who have BMI > or = 25 and <30.
- Obese women: Women with implant for more than twelve months who have BMI > or = 30.

SUMMARY:
Two-thirds of young women in the United States are overweight or obese. This excess weight may affect how their body metabolizes drugs such as different birth control methods. There is a not a lot of research about how excess weight could affect the hormone levels of the contraceptive implant. Methods like the implant contain only progesterone, which is a hormone that does not increase a woman's risk of blood clot. These methods would be preferred for overweight and obese women because excess weight also increases a woman's risk of blood clot.

The investigators propose a study comparing blood hormone levels of women using the implant for at least twelve months and in all weight categories. The investigators hope to show that all women, regardless of weight, will have hormone levels high enough to prevent pregnancy.

DETAILED DESCRIPTION:
Two-thirds of reproductive-age women in the United States are either overweight or obese. Body composition may affect contraceptive hormone metabolism and possibly efficacy. Phase III studies to date included few women weighing more than 70 kilograms (134 of 923, 14.5%); there were no reported pregnancies in that group. Data about pregnancy rates for women in higher body mass index (BMI) categories using the etonogestrel implant exists, but we know little about how weight affects the serum etonogestrel levels. Progestin-only methods, such as the etonogestrel implant, may be preferred over combined methods including estrogens because obesity increases thrombosis risk.

The investigators propose a prospective study to compare serum etonogestrel levels in the second and third years of implant use between women across body mass index categories.

Based on previous studies, the investigators expect a difference in etonogestrel levels based on body weight; however, the investigators hypothesize that etonogestrel levels will remain above the threshold for ovulation suppression through three years of implant use for women across BMI categories.

The investigators will measure the serum levels of etonogestrel in normal weight (BMI < 25kg/m2), overweight (BMI ≥ 25kg/m2 and < 30kg/m2), and obese women (BMI ≥ 30kg/m2) using the single-rod contraceptive implant for at least twelve months. Their primary objective is to compare the three groups and to evaluate whether etonogestrel levels fall below the critical level for contraceptive efficacy (90 pg/mL) (Díaz 1991) in any group.

ELIGIBILITY:
Inclusion Criteria:

* Woman using contraceptive implant for more than 12 months
* English or Spanish-speaking

Exclusion Criteria:

* None

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: The study population is English or Spanish-speaking women ages 15-45 years old at the New York Presbyterian Hospital's Title X Family Planning Clinic and the Columbia University Medical Center's Department of Obstetrics and Gynecology Family Planning Practice who have been using the etonogestrel contraceptive implant for at least the six months prior to their visit.
Sampling Method: Non-Probability Sample
Enrollment: 52 (Actual)
Dates: Start 2012-12; Primary Completion 2013-11 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
Serum Etonogestrel Level | Up to 12 months
  The investigators will measure the serum levels of etonogestrel in normal weight (BMI < 25kg/m2), overweight (BMI ≥ 25kg/m2 and < 30kg/m2), and obese women (BMI ≥ 30kg/m2) using the single-rod contraceptive implant for at least twelve months. The primary objective is to compare the three groups and to evaluate whether etonogestrel levels fall below the critical level for contraceptive efficacy (90 pg/mL) (Díaz 1991) in any group.

CONTACTS AND LOCATIONS:
Overall Officials: Kathleen M Morrell, MD, Principal Investigator — Columbia University
Locations (1):
- Columbia University Medical Center, New York, New York, United States

REFERENCES:
- [Background] Jacobson JC, Aikins Murphy P. United States medical eligibility criteria for contraceptive use 2010: a review of changes. J Midwifery Womens Health. 2011 Nov-Dec;56(6):598-607. doi: 10.1111/j.1542-2011.2011.00093.x. Epub 2011 Oct 17. PMID 22060220
- [Background] Ciangura C, Corigliano N, Basdevant A, Mouly S, Decleves X, Touraine P, Lloret-Linares C. Etonorgestrel concentrations in morbidly obese women following Roux-en-Y gastric bypass surgery: three case reports. Contraception. 2011 Dec;84(6):649-51. doi: 10.1016/j.contraception.2011.03.015. Epub 2011 May 8. PMID 22078197
- [Background] Davies GC, Feng LX, Newton JR, Van Beek A, Coelingh-Bennink HJ. Release characteristics, ovarian activity and menstrual bleeding pattern with a single contraceptive implant releasing 3-ketodesogestrel. Contraception. 1993 Mar;47(3):251-61. doi: 10.1016/0010-7824(93)90042-6. PMID 8462316
- [Background] Diaz S, Pavez M, Moo-Young AJ, Bardin CW, Croxatto HB. Clinical trial with 3-keto-desogestrel subdermal implants. Contraception. 1991 Oct;44(4):393-408. doi: 10.1016/0010-7824(91)90030-j. PMID 1756627
- [Background] Graesslin O, Korver T. The contraceptive efficacy of Implanon: a review of clinical trials and marketing experience. Eur J Contracept Reprod Health Care. 2008 Jun;13 Suppl 1:4-12. doi: 10.1080/13625180801942754. PMID 18330813
- [Background] Flegal KM, Carroll MD, Kit BK, Ogden CL. Prevalence of obesity and trends in the distribution of body mass index among US adults, 1999-2010. JAMA. 2012 Feb 1;307(5):491-7. doi: 10.1001/jama.2012.39. Epub 2012 Jan 17. PMID 22253363
- [Background] Huber J, Wenzl R. RETRACTED: Pharmacokinetics of Implanon. An integrated analysis. Contraception. 1998 Dec;58(6 Suppl):85S-90S. doi: 10.1016/s0010-7824(98)00120-6. PMID 10095978 (Retraction: PMID 15504385 Rekers H, Affandi B. Contraception. 2004 Nov;70(5):433)
- [Background] Mornar S, Chan LN, Mistretta S, Neustadt A, Martins S, Gilliam M. Pharmacokinetics of the etonogestrel contraceptive implant in obese women. Am J Obstet Gynecol. 2012 Aug;207(2):110.e1-6. doi: 10.1016/j.ajog.2012.05.002. Epub 2012 May 8. PMID 22717269
- [Background] Schnabel P, Merki-Feld GS, Malvy A, Duijkers I, Mommers E, van den Heuvel MW. Bioequivalence and x-ray visibility of a radiopaque etonogestrel implant versus a non-radiopaque implant: a 3-year, randomized, double-blind study. Clin Drug Investig. 2012 Jun 1;32(6):413-22. doi: 10.2165/11631930-000000000-00000. PMID 22540269
- [Background] Sivin I, Wan L, Ranta S, Alvarez F, Brache V, Mishell DR Jr, Darney P, Biswas A, Diaz S, Kiriwat O, Anant MP, Klaisle C, Pavez M, Schechter J. Levonorgestrel concentrations during 7 years of continuous use of Jadelle contraceptive implants. Contraception. 2001 Jul;64(1):43-9. doi: 10.1016/s0010-7824(01)00226-8. PMID 11535213
- [Background] Xu H, Wade JA, Peipert JF, Zhao Q, Madden T, Secura GM. Contraceptive failure rates of etonogestrel subdermal implants in overweight and obese women. Obstet Gynecol. 2012 Jul;120(1):21-6. doi: 10.1097/AOG.0b013e318259565a. PMID 22678035
- [Derived] Morrell KM, Cremers S, Westhoff CL, Davis AR. Relationship between etonogestrel level and BMI in women using the contraceptive implant for more than 1 year. Contraception. 2016 Mar;93(3):263-5. doi: 10.1016/j.contraception.2015.11.005. Epub 2015 Nov 11. PMID 26577754
- See also: Nexplanon Prescribing information — http://www.merck.com/product/usa/pi_circulars/n/nexplanon/nexplanon_pi.pdf